CLINICAL TRIAL: NCT06404034
Title: Expanded Access to Gallium Maltolate (GaM) for Adult Patients With Relapsed/Refractory Histologic or Molecular Glioblastoma
Brief Title: Expanded Access to Gallium Maltolate (GaM)
Status: Available | Type: Expanded Access
Sponsor: Imaging Biometrics, LLC (Industry)
Collaborators: xCures (Industry)
Responsible Party: Sponsor
Other Study IDs: IB-EAP-100
Record Dates: First submitted 2024-05-02; First posted 2024-05-08 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Glioblastoma; Refractory Glioblastoma; Glioblastoma Multiforme
Keywords: glioblastoma; refractory glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — gallium maltolate

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Gallium Maltolate — GaM will be provided as 500 mg capsules and will be self-administered once daily by mouth at the assigned dose level on a 28-day cycle (one cycle is 28 days) on an empty stomach. GaM should be taken at least 60 minutes before a meal and at least two hours after a meal. Liquids are allowed
  Other Names: GaM

SUMMARY:
The objective of this program is to provide GaM for compassionate use in patients with relapsed/refractory histologic or molecular glioblastoma who have exhausted available treatments.

The population of this program is adult patients aged greater than or equal to 18 years with a diagnosis of relapsed/refractory histologic or molecular glioblastoma, according to the WHO 2021 diagnostic criteria.

Molecular glioblastoma is characterized as an IDH-wildtype diffuse and astrocytic glioma in adults if there is microvascular proliferation or necrosis or TERT promoter mutation or EGFR gene amplification or +7/-10 chromosome copy number changes

DETAILED DESCRIPTION:
This is an intermediate-sized expanded access treatment protocol. GaM (GaM) will be provided as 500 mg capsules and will be self-administered once daily by mouth at the assigned dose level on a 28-day cycle (one cycle is 28 days). Initially, the patients will be provided a three (3) cycle prescription (a 28-day supply with two refills); enough total supply of GaM for three full cycles to allow for self-administration at home. It should be taken on an empty stomach. After that initial period, subsequent GaM will be provided to patients for continued self-administration.

At the treating physician's discretion, additional medication(s) may be administered. Clinical use of cancer-supportive care therapies is unrestricted, but the non-emergent use of additional anti-cancer therapies requires prior consultation with xCures and Imaging Biometrics. xCures along with Imaging Biometrics will be consulted prior to the non-emergent administration of any additional anti-cancer medications. xCures, along with Imaging Biometrics, should be consulted prior to any schedule modifications or the addition of other therapy. The patients may discontinue therapy at any time for any reason. The treating physician can discontinue therapy with GaM at any time for any reason.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has relapsed/refractory histologic or molecular glioblastoma who, in the opinion of the treating physician, may benefit from treatment from GaM.
2. Male or female patient aged ≥ 18 years.
3. In the opinion of the treating physician, the patient has adequate organ function to tolerate GaM.
4. Patient must be able to swallow and retain orally administered medication.
5. For females of childbearing potential, negative urinary or serum pregnancy test.
6. Patients must be willing to highly effective contraception for both male and female patients throughout the treatment and for at least 4 months after last treatment administration.
7. Toxicities related to any prior treatments are either stable, stable on supportive therapy, resolved, or in the opinion of the treating physician, clinically non-significant.
8. Ability to understand a written informed consent document, and the willingness to sign it by the patient or legally authorized patient representative (LAR) or guardian.
9. Informed consent obtained for the XCELSIOR longitudinal outcomes registry (NCT03793088)

Exclusion Criteria:

1. Patient is already participating in or is able to enroll in a clinical trial of GaM.
2. Patient has received systemic therapy with an investigational agent within 5 half-lives or 14 days prior to starting GaM treatment, whichever is shorter.
3. Patients completing radiotherapy treatment less than 14 days prior to planned study treatment initiation.
4. Patient is taking oral iron supplements or iron chelators.
5. Current evidence of uncontrolled, significant intercurrent illness that would, in the treating physician's judgment, contraindicate the patient's treatment with GaM due to safety concerns.
6. Patients who, in the opinion of the treating physician, have not fully recovered from recent major surgery to a sufficient extent to tolerate treatment with GaM.
7. Known hypersensitivity to GaM or any component in its formulation.
8. Patients taking prohibited medications as described in the current Investigator's Brochure.
9. Patient is pregnant or actively breastfeeding

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Cancer Partners of Nebraska, Lincoln, Nebraska
  - Northwell Health, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina